CLINICAL TRIAL: NCT01761006
Title: A Single-Center Exploratory Study to Evaluate FeNO Using the NIOX MINO® Device in COPD Patients Aged ≥40 Years During and Following Recovery From an Acute COPD Exacerbation
Brief Title: Evaluation of FeNO During and Following Acute COPD Exacerbation
Status: Terminated | Type: Observational
Why Stopped: Study was activated initially. However, the necessary resources were not available to complete the research.
Sponsor: Wake Forest University (Other)
Collaborators: Aerocrine AB (Industry)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: IRB00021832
Record Dates: First submitted 2012-12-19; First posted 2013-01-04 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Exhaled Nitric Oxide; NIOX MINO; Acute COPD exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: NIOX MINO®

SUMMARY:
The purpose of this research study is to determine whether exhaled nitric oxide (FeNO) goes up during an acute exacerbation of Chronic Obstructive Pulmonary Disease (AECOPD) and whether the level of exhaled nitric oxide returns to normal in the weeks after an exacerbation.

DETAILED DESCRIPTION:
The purpose of this research study is to determine whether exhaled nitric oxide (FeNO) goes up during an acute exacerbation of COPD and whether the level of exhaled nitric oxide returns to normal in the weeks after an exacerbation. FeNO is measured with a medical device called the NIOX MINO®. The NIOX MINO® device has been cleared by the Food and Drug Administration (FDA) for use in children and adults age 7 and older to measure Fractional Exhaled Nitric Oxide (FeNO) in human breath.This information will be useful for determining whether FeNO may help predict the development of a COPD exacerbation and/or be useful for identifying patients who will have a beneficial therapeutic response to inhaled or systemic corticosteroids during a COPD exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 years and above, inclusive
* Sex: Males and Females
* Smoking History: ≥20 pack years.
* COPD Defined as an FEV1/ FVC or FEV1/SVC ratio <70% predicted.
* AECOPD defined as a clinically significant worsening of COPD symptoms requiring treatment with antibiotics and/or systemic steroids and/or hospitalization for same.

Exclusion Criteria:

* Use of Systemic Corticosteroids for more than 48 hours prior to Visit 1.
* AECOPD requiring mechanical ventilation
* Study Participation Outside of This Protocol: Patients currently enrolled in studies of Investigational or non-Investigational Drugs or Medical Devices and/or who participated in these studies within 30 days prior to this study are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected based on the fact that they are currently experiencing an acute COPD exacerbation. The study will be conducted at a single-center COPD Clinic at Wake Forest University Baptist Medical Center, Winston-Salem NC, USA. It is anticipated that approximately 35 Patients age 40 years and above will participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09-23 (Actual); Study Completion 2014-09-23 (Actual)

PRIMARY OUTCOMES:
Change in FeNO from Day 0 to the end of the study | Time points for measurement of the Primary Endpoint will be between Day 0 (considered baseline) and Visit 2/Day 14, Visit 3/Day 28 and Visit 4/Day 56.

SECONDARY OUTCOMES:
Change in FEV1/FVC from Day 0 to the end of the study | Time points for measurement of the Secondary Endpoints will be between Day 0 (considered baseline) and Visit 2/Day 14, Visit 3/Day 28 and Visit 4/Day 56.
  Secondary Endpoint: Change in proportion of a person's vital capacity that they are able to expire in the first second of expiration (FEV1/FVC)
Change in FEV1 from Day 0 to the end of the study | Time points for measurement of the Secondary Endpoints will be between Day 0 (considered baseline) and Visit 2/Day 14, Visit 3/Day 28 and Visit 4/Day 56.
  Secondary Endpoint: Change in Forced Expiratory Volume at one second (FEV1)
Change in FEF25-75 from Day 0 to the end of the study | Time points for measurement of the Secondary Endpoints will be between Day 0 (considered baseline) and Visit 2/Day 14, Visit 3/Day 28 and Visit 4/Day 56.
  Secondary Endpoint: Change in Forced Expiratory Flow at the 25% point to the 75% point (FEF25-75)
Change in PEF from Day 0 to the end of the study | Time points for measurement of the Secondary Endpoints will be between Day 0 (considered baseline) and Visit 2/Day 14, Visit 3/Day 28 and Visit 4/Day 56.
  Secondary Endpoint: Change in Peak Expiratory Flow (PEF)
Change in Inspiratory Capacity from Day 0 to the end of the study | Time points for measurement of the Secondary Endpoints will be between Day 0 (considered baseline) and Visit 2/Day 14, Visit 3/Day 28 and Visit 4/Day 56.
  Secondary Endpoint: Change in Inspiratory Capacity
Change in Slow Vital Capacity (SVC) from Day 0 to the end of the study | Time points for measurement of the Secondary Endpoints will be between Day 0 (considered baseline) and Visit 2/Day 14, Visit 3/Day 28 and Visit 4/Day 56.
  Secondary Endpoint: Change in Slow Vital Capacity
Change in FEV1/SVC from Day 0 to the end of the study | Time points for measurement of the Secondary Endpoints will be between Day 0 (considered baseline) and Visit 2/Day 14, Visit 3/Day 28 and Visit 4/Day 56.
  Secondary Endpoint: Change in the ratio of FEV1 to Slow Vital Capacity
Change in COPD Assessment Test (CAT) Responses from Day 0 to the end of the study | Time points for measurement of the Secondary Endpoints will be between Day 0 (considered baseline) and Visit 2/Day 14, Visit 3/Day 28 and Visit 4/Day 56.
  Secondary Endpoint: Change in the responses on the CAT

OTHER OUTCOMES:
Evaluation of FEV1/FVC, FEV1, FEF25-75, FEF50, PEF and Inspiratory Capacity By FeNO Level at Baseline | Time points for measurement of the Secondary Endpoints will be between Day 0 (considered baseline) and Visit 2/Day 14, Visit 3/Day 28 and Visit 4/Day 56.
  • Other endpoint - the secondary endpoints will be evaluated by FeNO level at baseline as follows:
  * FeNO ≤ 25 ppb versus FeNO > 25 ppb
  * FeNO <50 ppb versus FeNO ≥ 50 ppb
  * FeNO > 25 ppb and FeNO < 50 ppb versus FeNO<25 and versus FeNO ≥ 50 ppb

CONTACTS AND LOCATIONS:
Overall Officials: Jill Ohar, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806
- [Background] Barnes PJ, Dweik RA, Gelb AF, Gibson PG, George SC, Grasemann H, Pavord ID, Ratjen F, Silkoff PE, Taylor DR, Zamel N. Exhaled nitric oxide in pulmonary diseases: a comprehensive review. Chest. 2010 Sep;138(3):682-92. doi: 10.1378/chest.09-2090. PMID 20822990
- [Background] Centers for Disease Control and Prevention (CDC). Deaths from chronic obstructive pulmonary disease--United States, 2000-2005. MMWR Morb Mortal Wkly Rep. 2008 Nov 14;57(45):1229-32. PMID 19008792
- [Background] Dweik RA, Boggs PB, Erzurum SC, Irvin CG, Leigh MW, Lundberg JO, Olin AC, Plummer AL, Taylor DR; American Thoracic Society Committee on Interpretation of Exhaled Nitric Oxide Levels (FENO) for Clinical Applications. An official ATS clinical practice guideline: interpretation of exhaled nitric oxide levels (FENO) for clinical applications. Am J Respir Crit Care Med. 2011 Sep 1;184(5):602-15. doi: 10.1164/rccm.9120-11ST. PMID 21885636
- [Background] Miller JD, Foster T, Boulanger L, Chace M, Russell MW, Marton JP, Menzin J. Direct costs of COPD in the U.S.: an analysis of Medical Expenditure Panel Survey (MEPS) data. COPD. 2005 Sep;2(3):311-8. doi: 10.1080/15412550500218221. PMID 17146996
- [Background] Rennard SI. COPD: overview of definitions, epidemiology, and factors influencing its development. Chest. 1998 Apr;113(4 Suppl):235S-241S. doi: 10.1378/chest.113.4_supplement.235s. PMID 9552012
- [Background] Siva R, Green RH, Brightling CE, Shelley M, Hargadon B, McKenna S, Monteiro W, Berry M, Parker D, Wardlaw AJ, Pavord ID. Eosinophilic airway inflammation and exacerbations of COPD: a randomised controlled trial. Eur Respir J. 2007 May;29(5):906-13. doi: 10.1183/09031936.00146306. Epub 2007 Feb 14. PMID 17301099
- [Background] van den Toorn LM, Overbeek SE, de Jongste JC, Leman K, Hoogsteden HC, Prins JB. Airway inflammation is present during clinical remission of atopic asthma. Am J Respir Crit Care Med. 2001 Dec 1;164(11):2107-13. doi: 10.1164/ajrccm.164.11.2006165. PMID 11739143